CLINICAL TRIAL: NCT03667911
Title: Educational Virtual Reality Videos in Improving Bowel Preparation Quality and Satisfaction of Outpatients Intended for Colonoscopy: a Prospective Randomised Controlled Study
Brief Title: Virtual Reality Videos in Improving Bowel Preparation Quality of Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, DONG WU, Associate Professor of Gastroenterology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: ZS-1647
Record Dates: First submitted 2018-09-04; First posted 2018-09-12 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Patient Compliance; Colo-rectal Cancer
Keywords: bowel preparation; colonoscopy; virtual reality; patient education
MeSH Terms: conditions — Patient Compliance; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Only routine patient education on bowel preparation of colonoscopy. Give oral instructions on bowel preparation(including definition, significance, correct steps as well as dietary limitations) by a well-trained nurses or doctors. Written instructions are offered, which have the some contents.
- Virtual-reality Group (Experimental): Watch virtual reality videos after routine patient education(both oral and written instructions). Videos give instructions on correct steps of bowel preparation, points for attention, as well as actual images of bowel during colonoscopy in the case of both excellent and unsatisfactory bowel preparation.
  Interventions: Other: virtual reality videos

INTERVENTIONS:
Other: virtual reality videos — Watch virtual reality videos after routine patient education(both oral and written instructions). Videos give instructions on correct steps of bowel preparation, points for attention, as well as actual images of bowel during colonoscopy in the case of both excellent and unsatisfactory bowel preparation.
  Arms: Virtual-reality Group

SUMMARY:
Colonoscopy is the most important method to screen for colorectal cancer and precancerous lesions, whose efficacy is closely related with the quality of bowel preparation, requiring consuming purgatives and restricting the diet. Compliance to bowel preparation is highly dependent on patient education. In most cases, such education is offered only once at the time of colonoscopy scheduling by either oral or written instructions. However, about one in fourth patients still cannot achieve satisfactory bowel preparation quality. Various methods, including booklet, telephone or message reminders, smartphone applications, social media, online videos, have been used to aid patient education and prove effective. These methods can increase patient activation, which is an independent factor related to bowel preparation quality. Virtual reality(VR) videos are used in this study, giving patients direct impressions of colonoscopy. This study aims to explore whether VR videos can increase patient adherence and experience, as well as improve bowel preparation quality, compared with conventional patient education methods.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients indicated for elective colonoscopy: 1) For screening purposes: asymptomatic patients with average or high risk for colorectal cancer[1]; 2) For diagnostic purposes: patients presented with abnormal imaging or lower gastrointestinal symptoms including bloody stool, chronic diarrhea and abdominal pain[2].
* Never undergo colonoscopy before.
* Age 18-75 years.
* Written informed consent.

Exclusion Criteria:

* History of bowel surgery
* Comorbidity disorder (ascites, congestive heart failure, chronic renal failure, coronary vessel disease within the last 6 months)
* Drug use (eg, constipation drugs, laxatives, or anti-diarrheal agents)
* Pregnancy
* Severe constipation (<3 bowel movement/week)
* Inflammatory bowel disease
* Unable to watch VR videos (eg, blindness)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Boston bowel preparation score | During colonoscopy
  A 10-point scale assessing bowel preparation. A four-point scoring system applied to each of the three broad regions of the colon: the right colon (including the cecum and ascending colon), the transverse colon (including the hepatic and splenic flexures), and the left colon (including the descending colon, sigmoid colon, and rectum).
  0 = Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared.
  1. = Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid.
  2. = Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well.
  3. = Entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid. The wording of the scale was finalized after incorporating feedback from three colleagues experienced in colonoscopy.

SECONDARY OUTCOMES:
polyp detection rate (PDR) | During colonoscopy
  Proportion of patients found to have polyp, may be a quality indictor of colonoscopy
adenoma detection rate (ADR) | During colonoscopy
  Proportion of patients found to have adenoma, may be a quality indictor of colonoscopy
cecal intubation rate | During colonoscopy
  Proportion of passage of the colonoscope tip to a point proximal to the ileocecal valve, may be a quality indictor of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen G, Zhao Y, Xie F, Shi W, Yang Y, Yang A, Wu D. Educating Outpatients for Bowel Preparation Before Colonoscopy Using Conventional Methods vs Virtual Reality Videos Plus Conventional Methods: A Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2135576. doi: 10.1001/jamanetworkopen.2021.35576. PMID 34807255
- [Derived] Zhao Y, Xie F, Bai X, Yang A, Wu D. Educational virtual reality videos in improving bowel preparation quality and satisfaction of outpatients undergoing colonoscopy: protocol of a randomised controlled trial. BMJ Open. 2019 Aug 20;9(8):e029483. doi: 10.1136/bmjopen-2019-029483. PMID 31434774